CLINICAL TRIAL: NCT04522297
Title: Nor-epinephrine Versus Midodrine/Octreotide in Patients With Hepatorenal Acute Kidney Injury
Brief Title: Nor-epinephrine Versus Midodrine/Octreotide in Patients With Hepatorenal Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, Doaa abdelaziz, Lecturer of clinical pharmacy, National Hepatology & Tropical Medicine Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-2018
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Hepato-Renal Syndrome
MeSH Terms: conditions — Hepatorenal Syndrome | interventions — Midodrine; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midodrine/Octreotide (Experimental): oral midodrine plus octreotide as subcutaneous injection
  Interventions: Drug: Midodrine/Octreotide
- Nor-epinephrine (Active Comparator): Intravenous infusion norepinephrine
  Interventions: Drug: Nor-epinephrine

INTERVENTIONS:
Drug: Midodrine/Octreotide — oral midodrine plus octreotide as subcutaneous injection
  Other Names: albumin at doses of 20 to 40 g/day
  Arms: Midodrine/Octreotide
Drug: Nor-epinephrine — Intravenous infusion norepinephrine
  Other Names: albumin at doses of 20 to 40 g/day
  Arms: Nor-epinephrine

SUMMARY:
Hepatorenal syndrome is a functional renal impairment occurring in cirrhotic patients . It develops secondary to splanchnic arterial vasodilatation which decreases the effective blood volume, activate the renin-angiotensin-aldosterone system, and stimulate of sympathetic nervous system.This study aims to compare the efficacy of nor-epinephrine versus midodrine/ octreotide, together with intravenous albumin on renal functions of patients with hepatorenal acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

Both sexes aged 18 years or older having cirrhosis, ascites, and a diagnosis of HRS-AKI based on the 2015 International Club of Ascites (ICA) diagnostic criteria

Exclusion Criteria:

Serum creatinine (sCr) >7 mg/dL Hypotension (mean arterial pressure (MAP) <70 mm Hg) or sepsis. Recent treatment with vasopressors. Patients with severe cardiovascular disease Known allergy to study medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Full response | 10 days
  the proportion of patients achieved full response defined as return of serum creatinine to a value within 0.3 mg/dl of the baseline value

SECONDARY OUTCOMES:
Partial response | 10 days
  defined as a regression of at least one acute kidney injury stage with a fall in the serum creatinine value to ≥0.3 mg/dl above the baseline serum creatinine value
Reversal | 10 days
  Incidence of HRS reversal defined as at least one serum creatinine value of ≤ 1.5 mg/dl while on treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Abdelaziz yousef, Ph.D, Study Director — Fellow at The National Hepatology and Tropical Research medicine institute
Locations (1):
- The National Hepatology and Tropical Research medicine institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No